CLINICAL TRIAL: NCT00361582
Title: A Randomized, Double-Blind, Active- and Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Multiple Doses of CG5503 Immediate Release Formulation in Subjects Awaiting Primary Joint Replacement Surgery for End-Stage Joint Disease
Brief Title: A Study to Evaluate the Effectiveness and Safety of Multiple Doses of Tapentadol(CG5503) in Patients Awaiting Joint Replacement Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR011218
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2010-04

CONDITIONS: Osteoarthritis; Pain Assessment; Arthralgia
Keywords: Osteoarthritis; tapentadol; knee-replacement; hip replacement; pain
MeSH Terms: conditions — Osteoarthritis; Arthralgia; Pain | interventions — Tapentadol

INTERVENTIONS:
Drug: CG5503 IR; tapentadol

SUMMARY:
The purpose of this study is to evaluate in patients who are eligible for elective primary total or partial joint replacement of the hip or knee due to chronic osteoarthritis the efficacy (level of pain control) of CG5503 over 5 and 10 days compared with placebo, and to assess the safety and tolerability of multiple doses of CG5503 IR patients.

DETAILED DESCRIPTION:
CG5503 is a centrally active pain-relieving drug being investigated for the treatment of acute and chronic pain. This study was designed to assess the safety and tolerability of CG5503 IR in patients who need joint replacement of the hip or knee due to chronic osteoarthritis. This is a double-blind study, i.e., neither patients nor investigators will know what treatment is given. Before the start of the 10 day double-blind phase, each patient will be screened for eligibility and eligible patients will be randomly assigned to receive either CG5503 IR, oxycodone IR, or placebo (i.e., no active drug). All patients will take their treatment by mouth every 4 to 6 hours during waking hours. A total of 60 doses (up to 6 doses per day) of study treatment will be provided for each patient during the 10-day treatment phase. The study treatment will be dispensed on Day 1, and patients will take the first dose in the evening of the same day. The effectiveness of study treatment (CG5503 IR, oxycodone, or placebo) will be assessed using several measures, including 11 Point Pain Numerical Rating Scale, 5-Point Relief Numerical Rating Scale, and Patient Global Impression of Change. Using these scales, patients will indicate their pain intensity level, pain relief level, and overall status of their well-being. Safety and tolerability will be assessed using physical examination, monitoring of adverse events, clinical and laboratory measures, and 12 lead ECG results. The null hypothesis for the study is that all CG5503 IR dosage efficacy results are equal to placebo based on the 5-day SPID in the treatment of chronic pain caused by osteoarthritis. The alternative study hypothesis is that at least 1 CG5503 IR dose effect will be different from placebo effect. CG5503 IR 50 mg, 75 mg of the base, 10 mg oxycodone or placebo for 10 days taken by mouth every 4 to 6 hours during waking hours. Patients randomized to CG5503 IR 75 mg group will receive CG5503 IR 50 mg on Day 1 and 75 mg on Day 2 to 10. All doses of study treatment should be taken with approximately 120 mL of water with or with food.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic osteoarthritis of the hip or the knee based on clinical and radiographic (X-Ray) criteria defined by standard accepted guidelines
* candidate (qualifies) for primary one-sided total or partial joint replacement surgery due to noninflammatory, end-stage degenerative joint disease (arthritis)
* requires daily doses of analgesic medication for chronic pain.

Exclusion Criteria:

* History of seizure disorder or epilepsy suggested by the presence of any of the following
* History of chronic hepatitis B and C or human immunodeficiency virus, or presence of active hepatitis B and C within the past 3 months before screening
* currently treated with anticonvulsants, monoamine oxidase inhibitors, tricyclic antidepressant, neuroleptics, or serotonin norepinephrine reuptake inhibitors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome is the SPID (Sum of Pain Intensity Difference) calculated at 5 days.

SECONDARY OUTCOMES:
Secondary efficacy outcomes include, among others, the time to the first use of rescue medication, the distribution of responder rates, and the SPID over 2 and 10 days.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study to Evaluate the Effectiveness and Safety of Multiple Doses of Tapentadol(CG5503) in Patients Awaiting Joint Replacement Surgery — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=728&filename=CR011218_CSR.pdf